CLINICAL TRIAL: NCT06184542
Title: To Evaluate Safety and Preliminary Immunogenicity of the Diphtheria-Tetanus-acellular Pertussis Component Combined Vaccine in Children Aged 2 Months to 6 Years: A Randomized, Blinded, Active-controlled Phase I Clinical Trial
Brief Title: Phase I Clinical Trial of Diphtheria-Tetanus-acellular Pertussis Component Combined Vaccine
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Institute of Medical Biology, Chinese Academy of Medical Sciences (Other)
Collaborators: Sichuan Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 20200610
Record Dates: First submitted 2023-12-14; First posted 2023-12-28 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Diphtheria; Tetanus; Pertussis
MeSH Terms: conditions — Diphtheria; Tetanus; Whooping Cough | interventions — Immunization, Secondary; Pentavac

STUDY DESIGN:
Intervention Model Description: Three stages (Children, Toddlers, and Infants) will be conducted according to the age-escalating principle. If safety assessed by DSMB meets the criteria, then the enrollment of the next stage could be continued.
Who Masked: Participant
Masking Description: In this study, participants are blinded, and part of the investigators are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (11):
- Intervention (Children aged 6 years, one-dose) (Experimental): Diphtheria-Tetanus-acellular Pertussis Component Combined Vaccine in Children aged 6 years on Day 0
  Interventions: Biological: DTacP (one-dose booster)
- DT Control (Children aged 6 years, one-dose) (Active Comparator): Diphtheria-Tetanus Combined Vaccine in Children aged 6 years on Day 0
  Interventions: Biological: DT (one-dose booster)
- Intervention (Toddlers aged 18-24 months, one-dose) (Experimental): Diphtheria-Tetanus-acellular Pertussis Component Combined Vaccine in toddlers aged 18-24 months on Day 0
  Interventions: Biological: DTacP (one-dose booster)
- DTaP Control (Toddlers aged 18-24 months, one-dose) (Active Comparator): Diphtheria-Tetanus-acellular Pertussis Vaccine in toddlers aged 18-24 months on Day 0
  Interventions: Biological: DTaP (one-dose booster)
- PENTAXIM Control (Toddlers aged 18-24 months, one-dose) (Active Comparator): PENTAXIM (DTaP-IPV-Hib) Vaccine in toddlers aged 18-24 months on Day 0
  Interventions: Biological: PENTAXIM (one-dose booster)
- Intervention (Infants aged 3 months, three-dose) (Experimental): Diphtheria-Tetanus-acellular Pertussis Component Combined Vaccine in infants aged 3 months on an M3-M4-M5 immunization schedule
  Interventions: Biological: DTacP (three-dose primary vaccination)
- DTaP Control (Infants aged 3 months, three-dose) (Active Comparator): Diphtheria-Tetanus-acellular Pertussis Vaccine in infants aged 3 months on an M3-M4-M5 immunization schedule
  Interventions: Biological: DTaP (three-dose primary vaccination)
- PENTAXIM Control (Infants aged 3 months, three-dose) (Active Comparator): PENTAXIM (DTaP-IPV-Hib) Vaccine infants aged 3 months on an M3-M4-M5 immunization schedule
  Interventions: Biological: PENTAXIM (three-dose primary vaccination)
- Intervention (Infants aged 2 months, three-dose, 2-3-4) (Experimental): Diphtheria-Tetanus-acellular Pertussis Component Combined Vaccine in infants aged 2 months on an M2-M3-M4 immunization schedule
  Interventions: Biological: DTacP (three-dose primary vaccination)
- Intervention (Infants aged 2 months, three-dose, 2-4-6) (Experimental): Diphtheria-Tetanus-acellular Pertussis Component Combined Vaccine in infants aged 2 months on an M2-M4-M6 immunization schedule
  Interventions: Biological: DTacP (three-dose primary vaccination)
- PENTAXIM Control (Infants aged 2 months, three-dose) (Active Comparator): PENTAXIM (DTaP-IPV-Hib) Vaccine infants aged 2 months on an M2-M3-M4 immunization schedule
  Interventions: Biological: PENTAXIM (three-dose primary vaccination)

INTERVENTIONS:
Biological: DTacP (one-dose booster) — Diphtheria-Tetanus-acellular Pertussis Component Combined Vaccine of 0.5mL on Day 0
  Arms: Intervention (Children aged 6 years, one-dose); Intervention (Toddlers aged 18-24 months, one-dose)
Biological: DTacP (three-dose primary vaccination) — Diphtheria-Tetanus-acellular Pertussis Component Combined Vaccine of 0.5mL on the M3-M4-M5, M2-M3-M4, or M2-M4-M6 immunization schedule
  Arms: Intervention (Infants aged 2 months, three-dose, 2-3-4); Intervention (Infants aged 2 months, three-dose, 2-4-6); Intervention (Infants aged 3 months, three-dose)
Biological: DT (one-dose booster) — Diphtheria-Tetanus Combined Vaccine of 0.5mL on Day 0
  Arms: DT Control (Children aged 6 years, one-dose)
Biological: DTaP (one-dose booster) — Diphtheria-Tetanus-acellular Pertussis Vaccine of 0.5mL on Day 0
  Arms: DTaP Control (Toddlers aged 18-24 months, one-dose)
Biological: PENTAXIM (one-dose booster) — Diphtheria, Tetanus, acellular Pertussis, inactivated Polio, conjugate Haemophilus influenzae type b Combined Vaccine of 0.5mL on Day 0
  Arms: PENTAXIM Control (Toddlers aged 18-24 months, one-dose)
Biological: DTaP (three-dose primary vaccination) — Diphtheria-Tetanus-acellular Pertussis Vaccine of 0.5mL on an M3-M4-M5immunization schedule
  Arms: DTaP Control (Infants aged 3 months, three-dose)
Biological: PENTAXIM (three-dose primary vaccination) — Diphtheria, Tetanus, acellular Pertussis, inactivated Polio, conjugate Haemophilus influenzae type b Combined Vaccine of 0.5mL on the M3-M4-M5 or M2-M3-M4 immunization schedule
  Arms: PENTAXIM Control (Infants aged 2 months, three-dose); PENTAXIM Control (Infants aged 3 months, three-dose)

SUMMARY:
This study is a randomized, blinded, active-controlled phase I clinical trial to evaluate the safety and preliminary immunogenicity of the Diphtheria-Tetanus-acellular Pertussis Component Combined Vaccine (DTacP) in subjects (aged 2 months to 6 years). Primary safety endpoints are the occurrence of solicited adverse events within 30 minutes after each dose, the occurrence of solicited adverse events within 7 days after each dose, the occurrence of unsolicited adverse events within 30 days after each dose, and the occurrence of adverse events 30 days after immunization. The secondary safety endpoint is the occurrence of serious adverse events (SAEs) within 12 months after immunization. Secondary immunogenicity endpoints are the geometric mean concentration (GMC), geometric mean fold increase (GMFI), seropositive rates, seroconversion rates, or 4-fold increase rates of anti-DT, anti-TT, anti-PT, anti-FHA, and anti-PRN antibodies 30 days after immunization. The exploratory endpoints are the GMC, GMFI, seropositive rates, seroconversion rates, or 4-fold increase rates of anti-DT, anti-PT, and anti-FHA neutralizing antibodies 30 days after immunization in all groups, the GMC and seropositive rates of anti-DT, anti-TT, anti-PT, anti-FHA, and anti-PRN antibodies 12 months after primary immunization in the infant group, the seropositive rates and geometric mean tie (GMT) of anti- type I, type II, type III poliovirus neutralizing antibodies 30 days after immunization in all groups, the seropositive rates and geometric mean tie (GMT) of anti- type I, type II, type III poliovirus neutralizing antibodies 12 months after primary immunization in the infant group.

DETAILED DESCRIPTION:
This is a randomized, blinded, active-controlled phase I clinical trial to evaluate the safety and preliminary immunogenicity in 460 subjects (aged 2 months to 6 years). Then 40 children (aged 6 years), 60 toddlers (aged 18-24 months), and 360 infants (180 subjects aged 3 months and 180 subjects aged 2 months) are eligible for enrollment after assessing thorough medical history and physical examination according to the principle of age escalating from children to infants.

[First Stage] 40 Children (aged 6 years) in the first stage of the study will be randomly assigned to the vaccine cohort and DT cohort in a ratio of 1:1, that is, 20 subjects in such group will be injected with the DTacP vaccine while 20 subjects with the DT vaccine. All children will receive the injection in the deltoid muscle of the upper arm on Day 0. The safety evaluation will be conducted by the Data and Safety Monitoring Board (DSMB) through assessing the preliminary safety data between Day 0 and Day 7 after administration. If results given by DSMB meet the criterion (no more than 25% of participants experienced Grade 3 or above adverse events and/or laboratory abnormalities), the study will continue to the second stage.

[Second Stage] 60 Toddlers (aged 18-24 months) in the second stage of the study will be randomly assigned to the vaccine cohort, DTaP cohort, and Pentaxim cohort in a ratio of 1:1:1, that is, 20 subjects in such group will be injected with the DTacP vaccine, 20 subjects will be injected with the DTaP vaccine, and the 20 subjects will be injected with DTaP-IPV-Hib (Pentaxim). All toddlers will receive the injection in the deltoid muscle of the upper arm on Day 0. The safety evaluation will be conducted by the Data and Safety Monitoring Board (DSMB) through assessing the preliminary safety data between Day 0 and Day 7 after administration. If results given by DSMB meet the criterion (no more than 25% of participants experienced Grade 3 or above adverse events and/or laboratory abnormalities), the study will continue to the third stage.

[Third Stage] (1) 180 Children (aged 3 months) in the third stage of the study will be randomly assigned to the vaccine cohort, DTaP cohort, and Pentaxim cohort in a ratio of 1:1:1, that is, 60 subjects in such group will be injected with the DTacP vaccine, 60 subjects will be injected with the DTaP vaccine, and 60 subjects will be injected with DTaP-IPV-Hib (Pentaxim). The vaccine cohort will be randomly assigned to two sub-cohorts in a ratio of 1:1 according to different injection sites, that is, 30 subjects will receive three injections in the anterolateral midthigh while 30 subjects in the deltoid muscle of the upper arm on an M3-M4-M5 immunization schedule. The DTaP cohort will receive three injections in the deltoid muscle of the upper arm on an M3-M4-M5 immunization schedule. The Pentaxim cohort will receive three injections in the anterolateral midthigh on an M3-M4-M5 immunization schedule. (2) 180 Children (aged 2 months) in the third stage of the study will be randomly assigned to the vaccine cohort, and Pentaxim cohort in a ratio of 2:1, that is, 120 subjects in such group will be injected with the DTacP vaccine, and 60 subjects will be injected with DTaP-IPV-Hib (Pentaxim). The vaccine cohort will be randomly assigned to four sub-cohorts in a ratio of 1:1:1:1 according to different injection sites and immunization schedules, that is, 30 subjects will receive three injections in the anterolateral midthigh on an M2-M3-M4 immunization schedule, 30 subjects will receive three injections in the anterolateral midthigh on an M2-M4-M6 immunization schedule, 30 subjects will receive three injections in the deltoid muscle of the upper arm on an M2-M3-M4 immunization schedule, 30 subjects will receive three injections in the deltoid muscle of the upper arm on an M2-M4-M6 immunization schedule. The Pentaxim cohort will receive three injections in the anterolateral midthigh on an M2-M3-M4 immunization schedule.

The duration of children and toddlers for intervention is 1 day. Thus, the duration of each subject in these two groups will be approximately 12 months. The duration of infants for intervention is 2 or 4 months, and as infants will be followed up to 18 months old, thus, each subject in such group will be approximately 15 or 16 months.

For safety assessment, the observation and evaluation of adverse events from Day 0 to Day 30 after each dose will be conducted by diary/contact cards and investigators' phone calls. Besides, the observation and evaluation of serious adverse events up to 12 months after vaccination will be conducted by active reports by subjects' legal guardians, or investigators' phone calls as well as face-to-face visits. Meanwhile, subjects will be observed at the site for at least 30 minutes after each dose.

For laboratory examination, blood biochemistry, blood routine, and urine routine tests will be performed on Day 0 before vaccination as well as Day 4 after administration in Children and Toddlers groups. If one of these two groups meets the criteria assessed by DSMB that over 20% of subjects in each group experience grade 3 or above laboratory abnormalities related to investigational vaccines on Day 4, then blood biochemistry, blood routine, and urine routine tests will be performed in the Infant Group on Day 0 before first dose, Day 4 after first dose and Day 4 after third dose.

For immunogenicity assessment, antibodies against anti-DT, anti-TT, anti-PT, anti-FHA, and anti-PRN, as well as neutralizing antibodies against anti-DT, anti-PT, anti-FHA, and anti-type I, type II, and type III poliovirus will be assessed in all subjects before vaccination and 30 days after vaccination. Moreover, antibodies against anti-DT, anti-TT, anti-PT, anti-FHA, and anti-PRN, as well as neutralizing antibodies against anti-type I, type II, and type III poliovirus will be assessed in infants around 12 months after primary vaccination (aged 18 months).

ELIGIBILITY:
Inclusion Criteria:

* Age Requirement: children aged 6 years, toddlers aged 18-24 months, and infants aged 2-3 months at the time of enrollment
* Previous Vaccination Requirements: (a) Children (aged 6 years) enrolled in the study should have received four doses of the Diphtheria, Tetanus, and Pertussis combined vaccine, and not yet received the Diphtheria, Tetanus combined vaccine; (b) Toddlers (aged 18-24 months) enrolled in the study should have received three doses of Diphtheria, Tetanus, and Pertussis combined vaccine as well as three doses of the Polio vaccine, and not yet received the booster dose of Diphtheria, Tetanus, and Pertussis combined vaccine and the Polio vaccine; (c) Infants (aged 3 months) enrolled in the study should not have received diphtheria-tetanus-pertussis-containing vaccine, polio-containing vaccine, 13-valent pneumococcal polysaccharide conjugate vaccine, Haemophilus influenzae type b conjugate vaccine, or meningococcal group A and C polysaccharide conjugate vaccine; (d) Infants (aged 2 months) enrolled in the study should not received diphtheria-tetanus-pertussis-containing vaccine, polio-containing vaccine, 13-valent pneumococcal polysaccharide conjugate vaccine, or Haemophilus influenzae type b conjugate vaccine.
* Provision of Legal Identification: Volunteers and their legal guardians or appointed representatives must provide valid legal identification documents.
* Informed Consent: Legal guardians or appointed representatives of volunteers must have the capacity to understand the informed consent document and the research process, voluntarily participate, sign the informed consent form, and be able to comply with the requirements in the study as well as complete relevant visits on time.
* Birth Outcome Condition: Toddlers (aged 18-24 months) and Infants (aged 2-3 months) should be born at full term (37-42 weeks of gestation) with birth weight ≥2500g.
* Temperature Requirement: Axillary body temperature is no more than 37.3°C.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria will be not eligible for enrollment.

* Previous Diagnosis: Subjects diagnosed with pertussis, tetanus, or diphtheria disease.
* Special Conditions for Toddlers (aged 18-24 months) and Infants (aged 2-3 months): Subjects have been with abnormal labor (dystocia, instrumental delivery) or a history of asphyxia, nervous system damage, or clinically confirmed pathological jaundice.
* Allergic History: Subjects have a history of allergies to any component of the vaccine (such as aluminum hydroxide), or previous allergy or suspected allergy to any vaccine, or other serious adverse reactions, such as anaphylactic shock, laryngeal edema, anaphylactic purpura, thrombocytopenic purpura, local anaphylactic necrosis reaction, dyspnea, angioedema, systemic rash and/or urticaria.
* Vaccination History: Subjects received any inactivated vaccines or subunit vaccines within 7 days before vaccination (except COVID-19 vaccines) with the investigational vaccine, or any other live attenuated vaccines or COVID-19 vaccines within 14 days before vaccination
* Acute Illness: Subjects have acute illness (e.g., fever) or acute exacerbation of a chronic illness within 3 days before receipt of the first dose of the investigational vaccine
* Neurological and Mental Health: Subjects have a history or family history of seizures, epilepsy, and other encephalopathy and psychiatric disorders.
* Health Condition: Subjects have a major congenital malformation, developmental disability, or congenital disease (e.g., Down syndrome, sickle cell anemia, congenital neurological disorders), or other clinically diagnosed serious chronic disease, including but not limited to, serious diseases of the nervous system, cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal tract, respiratory system, metabolic system, skeletal system and other system and malignant tumor history.
* Blood Disease: Subjects have genetic bleeding tendency or coagulopathy, or a history of bleeding disorders.
* Infectious Disease: Subjects diagnosed with infectious diseases that may interfere with the study, such as tuberculosis, viral hepatitis, human immunodeficiency virus (HIV) infection, etc.
* Special Condition: Subjects who cannot tolerate venipuncture or have a history of needle and blood sickness.
* Organ Removal History: Subjects with surgical removal of the spleen or other vital organs for any reason.
* Blood Condition: Subjects with blood loss (≥400 ml) and receipt of blood or blood products in the 3 months before receipt of the first dose of the investigational vaccine
* Immune Therapy: Subjects received treatment with an immunosuppressive agent, such as long-term systemic glucocorticoid therapy (treatment with systemic glucocorticoids, such as prednisone or a similar agent, for more than 2 consecutive weeks within 6 months before receipt of the first dose of an investigational vaccine), except topical agents (such as ointments, eye drops, inhalers, or nasal sprays) that do not exceed the recommended dose in the label or have any signs of systemic exposure
* Participation in Other Clinical Studies: Subjects use any investigational or unregistered product (drug, biologic product, or device) within 3 months before receipt of the first dose of the investigational vaccine, plan to use such product during the duration of this study, or were enrolled in another clinical trial before enrollment in this study.
* Physical Examination: (a) Subjects with abnormal vital signs with clinical significance; (b) Subjects abnormal blood routine, blood biochemistry, and urine routine test indicators with clinical significance
* Investigator's Discretion: The final exclusion criterion is the investigator's discretion to determine whether a subject is suitable for participation in the study.

Contraindications of the second and third doses of the vaccine:

Subjects meeting any of the following contraindications will be not eligible for the following doses.

* Serious Adverse Events: Subjects experienced serious adverse events related to vaccination after the previous dose.
* Vaccination with other vaccines during the study: (a) Subjects received other diphtheria, Tetanus, and acellular pertussis combined vaccines except for the investigational vaccine after the previous dose during the study period; (b) Infants (C3 subgroup and D3 subgroup) received other polio vaccines after the previous dose during the study period.
* Ineligibility: Subjects cannot be eligible or meet exclusion criteria after the previous dose of the investigational vaccine, and the qualification should be determined by the investigator.
* Investigator's Discretion: Subjects determined by the investigator as unsuitable for the following study period.

Ages: 2 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 460 (Estimated)
Dates: Start 2023-12-23 (Actual); Primary Completion 2024-12-15 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Safety index-incidence of adverse events | 0-30 minutes after the first dose vaccination
  Incidence of adverse events after the first dose vaccination (Applicable for Infants)
Safety index-incidence of adverse events | 0-30 minutes after the second dose vaccination
  Incidence of adverse events after the second dose vaccination (Applicable for Infants)
Safety index-incidence of adverse events | 0-30 minutes after the third dose vaccination
  Incidence of adverse events after the third dose vaccination (Applicable for Infants)
Safety index-incidence of adverse events | 0-30 minutes after the booster dose
  Incidence of adverse events after the booster dose (Applicable for Toddlers and Children)
Safety index-incidence of solicited adverse events | Day 0 to 7 after the first dose vaccination
  Incidence of solicited adverse events after the first dose vaccination (Applicable for Infants)
Safety index-incidence of solicited adverse events | Day 0 to 7 after the second dose vaccination
  Incidence of solicited adverse events after the second dose vaccination (Applicable for Infants)
Safety index-incidence of solicited adverse events | Day 0 to 7 after the third dose vaccination
  Incidence of solicited adverse events after the third dose vaccination (Applicable for Infants)
Safety index-incidence of solicited adverse events | Day 0 to 7 after the booster dose
  Incidence of solicited adverse events after the booster dose (Applicable for Toddlers and Children)
Safety index-incidence of unsolicited adverse events | Day 0 to 30 after the first dose vaccination
  Incidence of unsolicited adverse events after the first dose vaccination (Applicable for Infants)
Safety index-incidence of unsolicited adverse events | Day 0 to 30 after the second dose vaccination
  Incidence of unsolicited adverse events after the second dose vaccination (Applicable for Infants)
Safety index-incidence of unsolicited adverse events | Day 0 to 30 after the third dose vaccination
  Incidence of unsolicited adverse events after the third dose vaccination (Applicable for Infants)
Safety index-incidence of unsolicited adverse events | Day 0 to 30 after the booster dose
  Incidence of unsolicited adverse events after the booster dose (Applicable for Toddlers and Children)
Safety index-incidence of adverse events | From the beginning of the vaccination up to 30 days after the last vaccination completed
  Occurrence of adverse events after vaccination

SECONDARY OUTCOMES:
Safety index-incidence of serious adverse events | From the beginning of the vaccination up to 12 months after the last vaccination completed
  Occurrence of serious adverse events after vaccination
Immunogenicity index-seroconversion or ≥4-fold increase rates of antibody against DT | Between baseline and Day 30 after vaccination
  Antibody assay will be performed using the ELISA method. Seroconversion will be defined as a change from seronegative (Antibody Concentration<0.1 IU/ml) to seropositive (Antibody Concentration≥0.1 IU/ml), or a ≥4-fold increase from baseline.
Immunogenicity index-seroconversion or ≥4-fold increase rates of antibody against TT | Between baseline and Day 30 after vaccination
  Antibody assay will be performed using the ELISA method. Seroconversion will be defined as a change from seronegative (Antibody Concentration<0.1 IU/ml) to seropositive (Antibody Concentration≥0.1 IU/ml), or a ≥4-fold increase from baseline.
Immunogenicity index-seroconversion or ≥4-fold increase rates of antibody against PT | Between baseline and Day 30 after vaccination
  Antibody assay will be performed using the ELISA method. Seroconversion will be defined as a change from seronegative (Antibody Concentration<20 IU/ml) to seropositive (Antibody Concentration≥20 IU/ml), or a ≥4-fold increase from baseline.
Immunogenicity index-seroconversion or ≥4-fold increase rates of antibody against FHA | Between baseline and Day 30 after vaccination
  Antibody assay will be performed using the ELISA method. Seroconversion will be defined as a change from seronegative (Antibody Concentration<20 IU/ml) to seropositive (Antibody Concentration≥20 IU/ml), or a ≥4-fold increase from baseline.
Immunogenicity index-seroconversion or ≥4-fold increase rates of antibody against PRN | Between baseline and Day 30 after vaccination
  Antibody assay will be performed using the ELISA method. Seroconversion will be defined as a change from seronegative (Antibody Concentration<20 IU/ml) to seropositive (Antibody Concentration≥20 IU/ml), or a ≥4-fold increase from baseline.
Immunogenicity index-geometric mean concentration (GMC) of antibody against DT | Day 30 after vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-geometric mean concentration (GMC) of antibody against TT | Day 30 after vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-geometric mean concentration (GMC) of antibody against PT | Day 30 after vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-geometric mean concentration (GMC) of antibody against FHA | Day 30 after vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-geometric mean concentration (GMC) of antibody against PRN | Day 30 after vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-geometric mean fold increase (GMFI) of antibody against DT | Between baseline and Day 30 after vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-geometric mean fold increase (GMFI) of antibody against TT | Between baseline and Day 30 after vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-geometric mean fold increase (GMFI) of antibody against PT | Between baseline and Day 30 after vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-geometric mean fold increase (GMFI) of antibody against FHA | Between baseline and Day 30 after vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-geometric mean fold increase (GMFI) of antibody against PRN | Between baseline and Day 30 after vaccination
  Antibody assay will be performed using the ELISA method
Immunogenicity index-seropositive rates of antibody against DT | Day 30 after vaccination
  Antibody assay will be performed using the ELISA method. Seropositive will be defined as the Antibody Concentration≥0.1 IU/ml.
Immunogenicity index-seropositive rates of antibody against TT | Day 30 after vaccination
  Antibody assay will be performed using the ELISA method. Seropositive will be defined as the Antibody Concentration≥0.1 IU/ml.
Immunogenicity index-seropositive rates of antibody against PT | Day 30 after vaccination
  Antibody assay will be performed using the ELISA method. Seropositive will be defined as the Antibody Concentration≥20 IU/ml.
Immunogenicity index-seropositive rates of antibody against FHA | Day 30 after vaccination
  Antibody assay will be performed using the ELISA method. Seropositive will be defined as the Antibody Concentration≥20 IU/ml.
Immunogenicity index-seropositive rates of antibody against PRN | Day 30 after vaccination
  Antibody assay will be performed using the ELISA method. Seropositive will be defined as the Antibody Concentration≥20 IU/ml.

OTHER OUTCOMES:
Immunogenicity index-seropositive rates of neutralizing antibody against DT | Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method. Seropositive will be defined as the antibody titer ≥ 1:4.
Immunogenicity index-seropositive rates of neutralizing antibody against PT | Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method. Seropositive will be defined as the antibody titer ≥ 1:4.
Immunogenicity index-seropositive rates of neutralizing antibody against FHA | Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method. Seropositive will be defined as the antibody titer ≥ 1:4.
Immunogenicity index-geometric mean titer (GMT) of neutralizing antibody against DT | Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method.
Immunogenicity index-geometric mean titer (GMT) of neutralizing antibody against PT | Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method.
Immunogenicity index-geometric mean titer (GMT) of neutralizing antibody against FHA | Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method.
Immunogenicity index-geometric mean fold increase (GMFI) of neutralizing antibody against DT | Between baseline and Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method.
Immunogenicity index-geometric mean fold increase (GMFI) of neutralizing antibody against PT | Between baseline and Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method.
Immunogenicity index-geometric mean fold increase (GMFI) of neutralizing antibody against FHA | Between baseline and Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method.
Immunogenicity index-seroconversion or ≥4-fold increase rates of neutralizing antibody against DT | Between baseline and Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method. Seroconversion will be defined as a change from seronegative (Antibody Concentration<0.1 IU/ml) to seropositive (≥ 1:4), or a ≥4-fold increase from baseline.
Immunogenicity index-seroconversion or ≥4-fold increase rates of neutralizing antibody against PT | Between baseline and Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method. Seroconversion will be defined as a change from seronegative (Antibody Concentration<0.1 IU/ml) to seropositive (≥ 1:4), or a ≥4-fold increase from baseline.
Immunogenicity index-seroconversion or ≥4-fold increase rates of neutralizing antibody against FHA | Between baseline and Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method. Seroconversion will be defined as a change from seronegative (Antibody Concentration<0.1 IU/ml) to seropositive (≥ 1:4), or a ≥4-fold increase from baseline.
Immunogenicity index-geometric mean concentration (GMC) of antibody against DT | 12 months after primary vaccination
  Antibody assay will be performed using the ELISA method. (Applicable for Infants)
Immunogenicity index-geometric mean concentration (GMC) of antibody against TT | 12 months after primary vaccination
  Antibody assay will be performed using the ELISA method. (Applicable for Infants)
Immunogenicity index-geometric mean concentration (GMC) of antibody against PT | 12 months after primary vaccination
  Antibody assay will be performed using the ELISA method. (Applicable for Infants)
Immunogenicity index-geometric mean concentration (GMC) of antibody against FHA | 12 months after primary vaccination
  Antibody assay will be performed using the ELISA method. (Applicable for Infants)
Immunogenicity index-geometric mean concentration (GMC) of antibody against PRN | 12 months after primary vaccination
  Antibody assay will be performed using the ELISA method. (Applicable for Infants)
Immunogenicity index-seropositive rates of antibody against DT | 12 months after primary vaccination
  Antibody assay will be performed using the ELISA method. Seropositive will be defined as the Antibody Concentration≥0.1 IU/ml. (Applicable for Infants)
Immunogenicity index-seropositive rates of antibody against TT | 12 months after primary vaccination
  Antibody assay will be performed using the ELISA method. Seropositive will be defined as the Antibody Concentration≥0.1 IU/ml. (Applicable for Infants)
Immunogenicity index-seropositive rates of antibody against PT | 12 months after primary vaccination
  Antibody assay will be performed using the ELISA method. Seropositive will be defined as the Antibody Concentration≥20 IU/ml. (Applicable for Infants)
Immunogenicity index-seropositive rates of antibody against FHA | 12 months after primary vaccination
  Antibody assay will be performed using the ELISA method. Seropositive will be defined as the Antibody Concentration≥20 IU/ml. (Applicable for Infants)
Immunogenicity index-seropositive rates of antibody against PRN | 12 months after primary vaccination
  Antibody assay will be performed using the ELISA method. Seropositive will be defined as the Antibody Concentration≥20 IU/ml. (Applicable for Infants)
Immunogenicity index-geometric mean titer (GMT) of neutralizing antibody against Type I Poliovirus | Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method.
Immunogenicity index-geometric mean titer (GMT) of neutralizing antibody against Type II Poliovirus | Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method.
Immunogenicity index-geometric mean titer (GMT) of neutralizing antibody against Type III Poliovirus | Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method.
Immunogenicity index-seropositive rate of neutralizing antibody against Type I Poliovirus | Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method. Seropositive will be defined as the antibody titer ≥ 1:8.
Immunogenicity index-seropositive rate of neutralizing antibody against Type II Poliovirus | Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method. Seropositive will be defined as the antibody titer ≥ 1:8.
Immunogenicity index-seropositive rate of neutralizing antibody against Type III Poliovirus | Day 30 after vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method. Seropositive will be defined as the antibody titer ≥ 1:8.
Immunogenicity index-geometric mean titer (GMT) of neutralizing antibody against Type I Poliovirus | 12 months after the primary vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method. (Applicable for Infants)
Immunogenicity index-geometric mean titer (GMT) of neutralizing antibody against Type II Poliovirus | 12 months after the primary vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method. (Applicable for Infants)
Immunogenicity index-geometric mean titer (GMT) of neutralizing antibody against Type III Poliovirus | 12 months after the primary vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method. (Applicable for Infants)
Immunogenicity index-seropositive rate of neutralizing antibody against Type I Poliovirus | 12 months after the primary vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method. Seropositive will be defined as the antibody titer ≥ 1:8. (Applicable for Infants)
Immunogenicity index-seropositive rate of neutralizing antibody against Type II Poliovirus | 12 months after the primary vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method. Seropositive will be defined as the antibody titer ≥ 1:8. (Applicable for Infants)
Immunogenicity index-seropositive rate of neutralizing antibody against Type III Poliovirus | 12 months after the primary vaccination
  Neutralizing antibody assay will be performed using the neutralization and ELISA method. Seropositive will be defined as the antibody titer ≥ 1:8. (Applicable for Infants)

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Dazhu Center for Disease Prevention and Control, Dazhou, Sichuan
  - Cuiping Center for Disease Prevention and Control, Yibin, Sichuan
  - Xingwen Center for Disease Prevention and Control, Yibin, Sichuan